CLINICAL TRIAL: NCT00383994
Title: Immunotherapy With NK Cell, Rituximab and Rhu-GMCSF in Non-Myeloablative Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0234; NCI-2012-01375 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Lymphoma; Leukemia; Transplantation, Stem Cell; Lymphoid Malignancies; Disorder Related to Transplantation
Keywords: Chronic Lymphocytic Leukemia; CLL; Non-Hodgkin's Lymphoma; B-Cell Lymphoma; Lymphoma; granulocyte-macrophage colony-stimulating factor; Leukemia; NK Cells; Rituximab; GM-CSF; Non-myeloablative Allogeneic Stem Cell Transplantation; Stem Cell Transplant
MeSH Terms: conditions — Lymphoma; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunotherapy with NK Cell, Rituximab + GM-CSF (Experimental): Immunotherapy in Non-myeloablative Allogeneic Stem Cell Transplantation
  GM-CSF = Granulocyte-Macrophage Colony-Stimulating Factor
  Interventions: Drug: GM-CSF; Drug: Rituximab; Biological: NK Cell Infusion

INTERVENTIONS:
Drug: GM-CSF — 250 micrograms subcutaneously 3 times a week for 4 weeks starting a day before the administration of Rituximab.
  Other Names: Sargramostim; Leukine
Drug: Rituximab — 375 mg/m^2 by vein followed by 1000 mg/m^2 weekly for 3 weeks for a total of 4 doses.
  Other Names: Rituxan
Biological: NK Cell Infusion — NK cells will be infused one week after the fourth dose of Rituximab and GM-CSF.

SUMMARY:
The goal of this clinical research study is to find out if giving a boost of natural killer (NK) cells from a donor combined with Rituxan (rituximab), can help to control disease in patients who have already received an allogeneic stem cell transplant. The safety of this treatment will also be studied. Participants have recurrent chronic lymphocytic leukemia (CLL) or lymphoma after non-myeloablative stem cell transplantation.

Primary Objectives:

1.0 To determine the safety of Natural Killer (NK) cells and Rituximab + rhu-Granulocyte-macrophage colony-stimulating factor (GMCSF) in patients with persistent or recurrent B-cell lymphoid malignancies after non-myeloablative stem cell transplantation.

2.0 To determine factors associated with response.

DETAILED DESCRIPTION:
Rituximab is designed to attach to lymphoma cells, causing them to die. GM-CSF and NK cells may increase rituximab's ability to kill these cells.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have your complete medical history recorded and a physical exam. Your blood (about 2 tablespoons) will be collected for routine tests. A bone marrow aspirate will be performed. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. You will have computerized tomography (CT) scans as well as positron emission tomography (PET) or gallium scans to learn the status of your disease. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found eligible to take part in this study, you will receive treatment as an outpatient. You will receive GM-CSF 3 times a week for 4 weeks through a vein, starting the day before you receive the administration of rituximab. You will receive rituximab over 4 to 8 hours through a vein, once weekly for 4 weeks. You will also get a boost of NK cells from the same donor from whom you received your original transplant. These cells will be infused through a vein (over 30 to 60 minutes) after the 4th dose of rituximab. If you are receiving a cell infusion from somebody who you are not related to, the infusion may have to be done later if cells were not available as scheduled.

The CliniMACS System is a medical device that is used to separate types of blood cells from blood that is removed from the body during leukapheresis. These separated cells are processed for use in treatments such as stem cell transplants.

During this treatment, you will be examined as needed, and blood samples (1 tablespoon once or twice a week) will be taken for routine tests. You may need to receive blood transfusions during this study if your blood cell counts remain low.

You may be taken off this study if your disease gets worse or intolerable side effects occur.

You will have long-term, follow-up visits while on study. You will be seen at 4 to 6 weeks after you receive NK cell infusion; every 3 months during the first year; and then once a year. During each of these visits, you will have CT and PET scans, a bone marrow biopsy, and blood drawn (about 4 teaspoons) to learn the status of your disease.

This is an investigational study. Rituximab and GM-CSF are FDA approved and commercially available. NK cells are authorized by the FDA for use in research only. Up to 40 participants will take part in this study. All will be enrolled at the University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previous diagnosis of CD20+ B-cell CLL and non-Hodgkin's lymphoma who have failed standard conventional chemotherapy, and who had persistent disease at 3 months, or progressive disease after non-myeloablative allogeneic transplantation.
2. Donor willingness to donate peripheral blood (same donor of the original transplant).
3. Negative Beta HCG in a woman with child bearing potential defined as not post-menopausal for 12 months or not previous surgical sterilization.

Exclusion Criteria:

1. Pregnancy or lactation
2. HIV , HTLV-I or hepatitis.
3. Active infection(s) >/= grade 3.
4. Severe active concomitant medical or psychiatric illness.
5. Concurrent active GVHD requiring tacrolimus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) for NK cells infusions after non-myeloablative transplantation for lymphoid malignancies | Evaluated for toxicity within 6 weeks of treatment
  Maximum tolerated dose (MTD) is the highest dose with 10 patients treated and 5 or fewer patients with DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org